CLINICAL TRIAL: NCT03215290
Title: Application of Trans-parenchymal Compressing Suture in Major Liver Resection to Decrease Cutting Surface Related Complication.
Brief Title: Trans-parenchymal Compressing Suture in Major Liver Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Lei Dou, Principle Investigator, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TJ-201206
Record Dates: First submitted 2017-06-29; First posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Liver Carcinoma Resectable

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans-parenchymal compressing suture (Experimental): TCS: After liver transection, check for active hemorrhage and visible sites of bile leakage of cutting surface by stainless gauze which covered up on the raw cutting surface for 5 minutes. For patients with any positive findings including bloodstain and (or) bile staining, the cutting surface was recognized as "not good" cutting surface and further trans-parenchymal compressing sutured, if possible, using a hepatic needle.
  Interventions: Procedure: TCS
- Exposed surface (ES) (No Intervention): 147 Patients with exposed surface (ES) were matched as control group. No TCS.

INTERVENTIONS:
Procedure: TCS — The cutting surface recognized as "not good" cutting surface was further trans-parenchymal compressing sutured, if possible, using a hepatic needle.
  Other Names: trans-parenchymal compressing suture
  Arms: Trans-parenchymal compressing suture

SUMMARY:
Non-anatomical liver resection with appropriate resection margin was regarded as a potential curative treatment for selected major hepatic carcinoma due to preserving maximal normal liver, especially in cirrhotic patients. But occurrence of cutting surface related complications become a main challenge.

DETAILED DESCRIPTION:
In order to better manage the cutting surface after liver resection, we further applied trans-parenchymal compressing suture to "not good" cutting surface in hope of decreasing cutting surface related complication. A majority of studies investigating cutting surface management are limited to non-surgical treatments, such as the application of hemostasis agents including fibrin sealants, oxidized cellulose, and absorbable gelatin sponge13-15 . But there is no consensus regarding the necessity of the hemostatic agent application to the liver cutting surface. Up to date, few studies investigate surgical suture management of the cutting surface in liver resection.

ELIGIBILITY:
Inclusion Criteria:

1. tumor size more than 5cm
2. non-anatomical liver resection;

Exclusion Criteria:

1. intravascular infiltration with tumor embolus;
2. previous liver surgical treatment (e.g. microwave ablation; preoperative transcatheter arterial chemoembolization (TACE);
3. other concomitant extrahepatic procedures (e.g. splenectomy).
4. exposed Glisson Shealth, main hepatic veins or (and) retro-hepatic inferior vena cava.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Cutting surface related complications | 90 days
  After liver resection, some complication related cutting surface may occur, including surgery site infection, bile leakage, bleeding.

SECONDARY OUTCOMES:
Interventions for cutting surface related complications | 90 days
  Once the cutting surface related complications occur, some interventions need to be performed to treat these complications, such as percutaneous abdominal paracentesis or reoperation.